CLINICAL TRIAL: NCT00236015
Title: A 10-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Gabitril at 4, 8, and 12 mg/Day in the Treatment of Adults With Generalized Anxiety Disorder.
Brief Title: A 10-Week Efficacy and Safety Study of Gabitril in the Treatment of Adults With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: C6671/3030/AX/US
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders | interventions — Tiagabine

INTERVENTIONS:
Drug: Gabitril

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of an investigational anti-anxiety medication relative to placebo in patients with generalized anxiety disorder (GAD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 64 years of age (inclusive) will be eligible to participate if they satisfy the DSM-IV-TR criteria for GAD, as well as meeting the required screening and baseline visit scores for a series of psychiatric evaluations (i.e., HAM-A, HADS, MADRS and CGI-S).

Exclusion Criteria:

* Have been previously unresponsive to two or more adequate courses of pharmacological treatment for GAD
* Have been diagnosed with any other psychiatric Axis I disorder (except GAD) as a principal diagnosis within the past six months
* Have been diagnosed with any eating disorder within the past six months
* Have any history of OCD, psychotic disorder, bipolar disorder or antisocial personality disorder
* Have any history of alcohol or substance abuse within 3 months of screening
* Have any history of seizures, including febrile seizures
* Have any history of head trauma associated with loss of consciousness within the past 15 years

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 880
Dates: Start 2004-11; Study Completion 2006-03

PRIMARY OUTCOMES:
Reduction of symptomatology associated with Generalized Anxiety Disorder as assessed by the change from baseline to end point in the total score of the HAM-A scale.

SECONDARY OUTCOMES:
Assessment of proportion of responders and patients in remission according to HAM-A scores and CGI ratings by visit, assessment of the safety and tolerability in patients with GAD

CONTACTS AND LOCATIONS:
Locations (54):
- United States (48):
  - Pivotol Research Centers, Mesa, Arizona
  - Pivotal Research Center, Peoria, Arizona
  - Valley Clinical Research, El Centro, California
  - Radiant Research Irvine, Irvine, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Riverside, California
  - Clinical Innovations, Inc., Santa Ana, California
  - Radiant Research, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Miami Research Associates, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Roskamp Institute, Clinical Trials Division, Sarasota, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - American Medical Research, Aurora, Illinois
  - Henry Lahmeyer MD & Associates, Northfield, Illinois
  - Midwest Center for Neurobehavioral Medicine, Oakbrook Terrace, Illinois
  - Indiana University Hospital AOC, Indianapolis, Indiana
  - Vince & Associates Clinical Research, Overland Park, Kansas
  - Pedia Research, LLC, Owensboro, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - LSU Health Science Center, Shreveport, Louisiana
  - Capital Clinical Research Associates, Rockville, Maryland
  - Dupont Clinical Research, Rockville, Maryland
  - Center for Psychopharmacologic Research and Treatment, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Regions Hospital - Department of Behavioral Health, Saint Paul, Minnesota
  - Radiant Research, Las Vegas, Nevada
  - Center for Emotional Fitness, Moorestown, New Jersey
  - Fieve Clinical Services, Inc., New York, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - Medark Clinical Trials and Research, Morganton, North Carolina
  - Richard Weisler, MD and Associates, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - Pahl Pharmaceutical Research, LLC, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Eugene, Oregon
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - CNS Research Institute, Philadelphia, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Future Search Trials, Austin, Texas
  - Claghorn-Lesem Research Clinic, Inc., Bellaire, Texas
  - Mood Disorders Research Clinic; UT Southwestern Medical Center at Dallas, Dallas, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Croft Group Research Center, San Antonio, Texas
  - University of Utah Mood Disorders Clinic, Salt Lake City, Utah
  - Dean Foundation, Middleton, Wisconsin
- Canada (6):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Mood Disorders Clinic, Hamilton, Ontario
  - Center for Addiction and Mental Health, Mood and Anxiety Program, Toronto, Ontario
  - Clinique Marie-Fitzbach,, Québec, Quebec